CLINICAL TRIAL: NCT02435680
Title: A Randomized Phase II Study of MCS110 Combined With Carboplatin and Gemcitabine in Advanced Triple Negative Breast Cancer (TNBC)
Brief Title: Efficacy Study of MCS110 Given With Carboplatin and Gemcitabine in Advanced Triple Negative Breast Cancer (TNBC)
Acronym: TNBC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMCS110Z2201; 2015-000179-29 (EudraCT Number)
Record Dates: First submitted 2015-04-22; First posted 2015-05-06 (Estimated); Results first posted 2021-06-21 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-05

CONDITIONS: Advanced Triple Negative Breast Cancer (TNBC) With High TAMs
Keywords: MCS110; carboplatin; gemcitabine; TNBC; TAMs
MeSH Terms: interventions — Carboplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1: MCS110+carboplatin+gemcitabine (Experimental): MCS110+carboplatin+gemcitabine
  Interventions: Drug: MCS110; Drug: carboplatin; Drug: gemcitabine
- Arm 2: carboplatin+gemcitabine (Active Comparator): carboplatin+gemcitabine
  Interventions: Drug: carboplatin; Drug: gemcitabine

INTERVENTIONS:
Drug: MCS110 — taken by I.V
  Arms: Arm 1: MCS110+carboplatin+gemcitabine
Drug: carboplatin — taken by I.V
Drug: gemcitabine — taken by I.V

SUMMARY:
To determine whether MCS110 antibody therapy improves the efficacy of carboplatin and gemcitabine (carbo/gem) in advanced TNBC patients

ELIGIBILITY:
Inclusion Criteria:

* Adult women (≥ 18 years of age) with advanced TNBC.
* Histological or cytological evidence of estrogen-receptor negative (ER-), progesterone receptor negative (PgR-) and human epidermal growth factor-2 receptor negative (HER2-) Breast Cancer by local laboratory testing, based on last available tumor tissue.
* ER/PgR negativity to follow local guidelines
* If IHC HER2 2+, a negative FISH test is required
* A pre-treatment tumor biopsy demonstrating high TAM content as assessed per the central laboratory
* Patients must have:

At least one measurable lesion per RECIST 1.1. (Note: Measurable lesions include lytic or mixed (lytic + blastic) bone lesions, with an identifiable soft tissue component that meets the measurability criteria)

Exclusion Criteria:

* Prior chemotherapy for advanced BC. Previous adjuvant/neoadjuvant chemotherapy is allowed (carboplatin, cisplatin or gemcitabine only if > 12 months has passed since last administration).
* Therapy for underlying malignancy within 2 weeks prior to start of study treatment:
* Chemotherapy, biologic therapy (antibodies and biologically targeted small molecules)
* Radiotherapy
* Major surgery
* Patients receiving concomitant immunosuppressive agents or chronic corticosteroids (≥10 mg of prednisone or equivalent) at the time of first study dose.
* Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of screening.
* Known history of human immunodeficiency virus or active infection with hepatitis virus or any uncontrolled active systemic infection.
* Patients with the following laboratory values during screening and on Day 1 predose:
* Absolute Neutrophil Count (ANC) < 1.5x109/L
* Hemoglobin < 9 g/dL
* Platelets < 100x109/L
* Serum creatinine > 1.5 x ULN
* Serum total bilirubin > 1.5 x ULN
* AST/SGOT and ALT/SGPT > 3.0 x ULN

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-08-10 (Actual); Primary Completion 2020-01-04 (Actual); Study Completion 2020-03-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (22):
- United States (2):
  - Highlands Oncology Group, Fayetteville, Arkansas
  - Massachusetts General Hospital Cancer Center SC, Boston, Massachusetts
- Novartis Investigative Site, Nedlands, Western Australia, Australia
- Austria (2):
  - Novartis Investigative Site, Salzburg
  - Novartis Investigative Site, Vienna
- Novartis Investigative Site, Brussels, Belgium
- France (2):
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Saint-Herblain Cédex
- Germany (3):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Essen
- Novartis Investigative Site, Hong Kong SAR, Hong Kong
- Italy (2):
  - Novartis Investigative Site, Bologna
  - Novartis Investigative Site, Napoli
- South Korea (2):
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Seoul
- Spain (4):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Santiago de Compostela, Galicia
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
- Novartis Investigative Site, Taipei, Taiwan
- Novartis Investigative Site, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In total, 50 subjects were enrolled into the study and 49 subjects received study treatment.
Groups:
- MCS110+Carboplatin+Gemcitabine: experimental. MCS110 10mg/kg intravenous infusion on day 1.
- MCS110 With C1D8 Dose+Carboplatin+Gemcitabine: experimental.MCS110 10mg/kg intravenous infusion on day 1 and day 8
- Carboplatin+Gemcitabine: comparator. Gemcitabine: Intravenous infusion 1000 mg/m2 Days 1 & 8 Carboplatin: Intravenous infusion AUC 2 Days 1 & 8
Period: Overall Study
Arm/Group | MCS110+Carboplatin+Gemcitabine | MCS110 With C1D8 Dose+Carboplatin+Gemcitabine | Carboplatin+Gemcitabine
Started | 21 | 13 | 16
Completed | 0 | 0 | 0
Not Completed | 21 | 13 | 16
Not completed — Physician Decision | 3 | 0 | 0
Not completed — subject / guardian decision | 0 | 3 | 2
Not completed — Adverse Event | 8 | 3 | 2
Not completed — progressive disease | 10 | 7 | 11
Not completed — not treated | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- MCS110 With C1D8 Dose + Carboplatin +Gemcitabine: experimental.MCS110 10mg/kg intravenous infusion on days 1 & 8
- Total: Total of all reporting groups
Arm/Group | MCS110+Carboplatin+Gemcitabine | MCS110 With C1D8 Dose + Carboplatin +Gemcitabine | Carboplatin+Gemcitabine | Total
Number analyzed (Participants) | 21 | 13 | 16 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.5 (13.20) | 56.2 (12.97) | 55.1 (13.20) | 55.5 (12.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 13 | 16 | 50
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 15 | 10 | 11 | 36
  Asian | 2 | 2 | 3 | 7
  Unknown | 3 | 1 | 1 | 5
  Other | 1 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) as Per RECIST v1.1 (by Local Investigator Assessment)
Description: PFS Results presented for all MCS110 treated patients (with and without day 8 dose), in line with phase 2 study design.
Time Frame: 4 years
Population: full analysis set: all MCS110 treated patients versus comparator
Measure: Median (90% Confidence Interval); unit: months
Groups:
- All MCS110+Carboplatin+Gemcitabine: experimental. all MCS110 treated patients, with 10mg/kg intravenous infusion, on day 1 and days 1 & 8
Arm/Group | All MCS110+Carboplatin+Gemcitabine | Carboplatin+Gemcitabine
Number analyzed (Participants) | 34 | 16
months | 5.6 [4.5 to 8.7] | 5.5 [3.5 to 7.5]

2. Secondary Outcome: Free MCS110 : Derived Pharmacokinetics (PK) Parameters: AUCtau
Description: AUC tau derived from day 0 to 21 (cycle 1) from day 0 to 21 (cycle 4) Cycle duration is 21 days
Time Frame: day 21 (end cycle 1); day 84 (end cycle 4)
Population: pharmacokinetic analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day * microgram / mL
Arm/Group | MCS110+Carboplatin+Gemcitabine | MCS110 With C1D8 Dose + Carboplatin +Gemcitabine
Number analyzed (Participants) | 19 | 15
day * microgram / mL
  day 21: number analyzed (Participants) | 17 | 9
  day 21 | 1430 (23.5) | 2960 (22.7)
  day 84: number analyzed (Participants) | 8 | 2
  day 84 | 1840 (34.9) | 3240 (30.0)

3. Secondary Outcome: Free MCS110 : Derived Pharmacokinetics (PK) Parameters: Cmax
Time Frame: day 21 (end cycle 1); day 84 (end cycle 4)
Population: pharmacokinetic analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram / mL
Arm/Group | MCS110+Carboplatin+Gemcitabine | MCS110 With C1D8 Dose + Carboplatin +Gemcitabine
Number analyzed (Participants) | 19 | 15
microgram / mL
  day 21: number analyzed (Participants) | 18 | 12
  day 21 | 186 (28.5) | 281 (21.2)
  day 84: number analyzed (Participants) | 9 | 2
  day 84 | 240 (14.8) | 319 (27.8)

4. Secondary Outcome: Cmax Derived From Plasma Concentration of Carboplatin, Gemcitabine and 2',2'-Difluoro-deoxyuridine (dFdU)
Description: day 21 (end cycle 1); day 84 (end cycle 4)
Time Frame: day 21, day 84
Population: pharmacokinetic analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram /mL
Arm/Group | MCS110+Carboplatin+Gemcitabine | MCS110 With C1D8 Dose + Carboplatin +Gemcitabine | Carboplatin+Gemcitabine
Number analyzed (Participants) | 19 | 15 | 15
nanogram /mL
  Cmax Carboplatin Day 21: number analyzed (Participants) | 16 | 13 | 14
  Cmax Carboplatin Day 21 | 12400 (37.3) | 12500 (33.2) | 11200 (70.9)
  Cmax Carboplatin Day 84: number analyzed (Participants) | 11 | 6 | 10
  Cmax Carboplatin Day 84 | 9550 (33.0) | 10000 (28.9) | 11600 (55.0)
  Cmax Gemcitabine Day 21: number analyzed (Participants) | 16 | 13 | 13
  Cmax Gemcitabine Day 21 | 2750 (194.5) | 5480 (95.1) | 2370 (484.9)
  Cmax Gemcitabine Day 84: number analyzed (Participants) | 12 | 6 | 9
  Cmax Gemcitabine Day 84 | 2470 (227.3) | 3400 (173.9) | 8630 (101.2)
  Cmax dFdU Day 21: number analyzed (Participants) | 16 | 13 | 13
  Cmax dFdU Day 21 | 39100 (21.6) | 33900 (19.5) | 37700 (28.2)
  Cmax dFdU Day 84: number analyzed (Participants) | 13 | 6 | 9
  Cmax dFdU Day 84 | 36600 (88.6) | 30300 (11.8) | 32300 (12.4)

5. Secondary Outcome: AUClast Derived From Plasma Concentration of Carboplatin, Gemcitabine and 2',2'-Difluoro-deoxyuridine (dFdU)
Description: day 21 (end cycle 1); day 84 (end cycle 4)
Time Frame: day 21, day 84
Population: pharmacokinetic analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours * nanogram /mL
Arm/Group | MCS110+Carboplatin+Gemcitabine | MCS110 With C1D8 Dose + Carboplatin +Gemcitabine | Carboplatin+Gemcitabine
Number analyzed (Participants) | 19 | 15 | 15
hours * nanogram /mL
  AUC Carboplatin Day 21: number analyzed (Participants) | 16 | 13 | 14
  AUC Carboplatin Day 21 | 24500 (31.1) | 21400 (27.3) | 21800 (56.0)
  AUC Carboplatin Day 84: number analyzed (Participants) | 11 | 6 | 10
  AUC Carboplatin Day 84 | 18300 (21.8) | 17500 (25.0) | 20500 (34.6)
  AUC Gemcitabine Day 21: number analyzed (Participants) | 16 | 13 | 13
  AUC Gemcitabine Day 21 | 2390 (157.3) | 4270 (79.3) | 2620 (225.5)
  AUC Gemcitabine Day 84: number analyzed (Participants) | 12 | 6 | 9
  AUC Gemcitabine Day 84 | 2410 (115.2) | 2770 (118.8) | 6320 (76.2)
  AUC dFdU Day 21: number analyzed (Participants) | 16 | 13 | 13
  AUC dFdU Day 21 | 230000 (34.7) | 181000 (37.7) | 231000 (25.2)
  AUC dFdU Day 84: number analyzed (Participants) | 13 | 6 | 9
  AUC dFdU Day 84 | 229000 (31.9) | 147000 (28.7) | 211000 (24.7)

6. Secondary Outcome: Total Colony Stimulation Factor -1 (CSF-I) Circulating Levels
Description: results expressed as a the ratio change from baseline expressed in percentage. Cycle duration is 21 days. These Biomarker Analyses were performed for MCS110 treated patients only.
Time Frame: baseline, day 1, 4, 15, 22, 43, 64, 85, 106, 127, 148
Population: Safety set - MCS110 treated patients only
Measure: Mean (Standard Deviation); unit: % change from baseline
Arm/Group | MCS110+Carboplatin+Gemcitabine | MCS110 With C1D8 Dose + Carboplatin +Gemcitabine
Number analyzed (Participants) | 19 | 15
% change from baseline
  Day 1: number analyzed (Participants) | 16 | 13
  Day 1 | 110 (19.8) | 115 (34.8)
  Day 4: number analyzed (Participants) | 10 | 9
  Day 4 | 4930 (2280) | 4350 (1620)
  Day 15: number analyzed (Participants) | 17 | 13
  Day 15 | 21600 (8290) | 19500 (6130)
  Day 22 (cycle 2 day 1): number analyzed (Participants) | 15 | 8
  Day 22 (cycle 2 day 1) | 32000 (9190) | 34400 (14900)
  Day 43 (cycle 3 day 1): number analyzed (Participants) | 16 | 6
  Day 43 (cycle 3 day 1) | 57900 (14100) | 70000 (27400)
  Day 64 (cycle 4 day 1): number analyzed (Participants) | 11 | 5
  Day 64 (cycle 4 day 1) | 73600 (16200) | 78000 (41200)
  Day 85 (cycle 5 day 1): number analyzed (Participants) | 9 | 4
  Day 85 (cycle 5 day 1) | 79300 (27000) | 107000 (51400)
  Day 106 (cycle 6 day 1): number analyzed (Participants) | 4 | 5
  Day 106 (cycle 6 day 1) | 97500 (15600) | 103000 (50700)
  Day 127 (cycle 7 day 1): number analyzed (Participants) | 3 | 5
  Day 127 (cycle 7 day 1) | 110000 (33800) | 109000 (40100)
  Day 148 (cycle 8 day 1): number analyzed (Participants) | 3 | 3
  Day 148 (cycle 8 day 1) | 108000 (30300) | 111000 (58800)

7. Secondary Outcome: Serum C-terminal Telopeptide of Type I Collagen (CTX-I)
Description: results expressed as a the ratio change from baseline expressed in percentage. Cycle duration is 21 days.
  Biomarker Analyses performed for MCS110 treated patients only.
Time Frame: baseline, day 2, 4, 15, 22, 43, 64, 85, 106, 127, 148
Population: Safety set - MCS110 treated patients only
Measure: Mean (Standard Deviation); unit: % change from baseline
Arm/Group | MCS110+Carboplatin+Gemcitabine | MCS110 With C1D8 Dose + Carboplatin +Gemcitabine
Number analyzed (Participants) | 19 | 15
% change from baseline
  Day 2: number analyzed (Participants) | 18 | 12
  Day 2 | 79.4 (22.8) | 85.0 (44.0)
  Day 4: number analyzed (Participants) | 15 | 11
  Day 4 | 72.5 (25.4) | 80.2 (39.6)
  Day 15: number analyzed (Participants) | 16 | 14
  Day 15 | 65.6 (44.3) | 69.4 (27.4)
  Day 22 (cycle 2 day 1): number analyzed (Participants) | 17 | 14
  Day 22 (cycle 2 day 1) | 67.9 (43.6) | 52.9 (26.5)
  Day 43 (cycle 3 day 1): number analyzed (Participants) | 17 | 8
  Day 43 (cycle 3 day 1) | 64.3 (58.7) | 39.3 (23.8)
  Day 64 (cycle 4 day 1): number analyzed (Participants) | 15 | 7
  Day 64 (cycle 4 day 1) | 69.7 (62.2) | 29.5 (23.7)
  Day 85 (cycle 5 day 1): number analyzed (Participants) | 11 | 7
  Day 85 (cycle 5 day 1) | 102 (124) | 40.6 (34.8)
  Day 106 (cycle 6 day 1): number analyzed (Participants) | 7 | 7
  Day 106 (cycle 6 day 1) | 41.2 (13.2) | 50.2 (45.3)
  Day 127 (cycle 7 day 1): number analyzed (Participants) | 4 | 5
  Day 127 (cycle 7 day 1) | 38.7 (14.9) | 68.7 (66.5)
  Day 148 (cycle 8 day 1): number analyzed (Participants) | 4 | 4
  Day 148 (cycle 8 day 1) | 40.5 (13.7) | 75.3 (103)

8. Secondary Outcome: Tumor Response Per RECIST v1.1 (by Local Investigator Assessment)
Description: CR: complete response. PR: partial response. SD: stable disease: CBR: clinical benefit rate =CR + PR + SD lasting at least for 6 months. ORR = CR + PR. Efficacy Results presented for all MCS110 treated patients (with and without day 8 dose), in line with phase 2 study design.
Time Frame: 4 years
Population: full analysis set: all MCS110 treated patients versus comparator
Measure: Count of Participants; unit: Participants
Arm/Group | MCS110+Carboplatin+Gemcitabine | Carboplatin+Gemcitabine
Number analyzed (Participants) | 34 | 16
Participants
  PR | 8 | 6
  Non-CR/ Non-progressive disease | 1 | 0
  SD | 19 | 7
  progressive disease | 4 | 1
  unknown | 2 | 2
  clinical benefit rate | 10 | 7
  ORR | 8 | 6

9. Secondary Outcome: Tumor Response Per RECIST v1.1 (by Local Investigator Assessment) Duration of Response
Description: as for outcome 8
Time Frame: 4 years
Population: full analysis set: all MCS110 treated patients versus comparator
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | MCS110+Carboplatin+Gemcitabine | Carboplatin+Gemcitabine
Number analyzed (Participants) | 34 | 16
months | 9.6 [3.6 to 42.5] | 5 [2.7 to 13.3]

10. Secondary Outcome: Number of Patients With at Least One MCS110 Dose Reduction, and Number of Patients With at Least One MCS110 Dose Interruption
Description: patients treated with MCS110 only
Time Frame: 4 years
Population: Safety set - MCS110 treated patients only
Measure: Count of Participants; unit: Participants
Arm/Group | MCS110+Carboplatin+Gemcitabine | MCS110 With C1D8 Dose + Carboplatin +Gemcitabine
Number analyzed (Participants) | 19 | 15
Participants
  MCS110 dose reduction | 3 | 5
  MCS110 dose interruption | 6 | 9

11. Secondary Outcome: MCS110 Dose Intensity
Description: Relative dose intensity by categories.
  Patients treated with MCS110 only. The dose intensity measures the dose actually taken versus the planned dose, and is expressed in percentage:
  <50%: less than 50 % of the planned dose received; 50-<75 %: dose received is 50% or more, but less than 75 %; 75-<90 %: dose received is 75% or more, but less than 90%; 90-<110 %: dose received is 90% or more, but less than 110%
Time Frame: 4 years
Population: Safety set - MCS110 treated patients only
Measure: Count of Participants; unit: Participants
Arm/Group | MCS110+Carboplatin+Gemcitabine | MCS110 With C1D8 Dose + Carboplatin +Gemcitabine
Number analyzed (Participants) | 19 | 15
Participants
  <50% | 1 | 4
  50-<75% | 8 | 3
  75-<90% | 7 | 5
  90-<110% | 3 | 3

12. Secondary Outcome: Tumor Associated Macrophage (TAM) and Tumor Infiltrating Lymphocyte (TIL) Content in Pre- and Post-dose Tumor Biopsies.
Description: results expressed as a the ratio change from baseline expressed in percentage: Biopsies were taken at baseline and between Day 29 and Day 43. Patients treated with MCS110 only
Time Frame: Baseline, Day 29-43
Population: Safety set - MCS110 treated patients only
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: % change from baseline
Arm/Group | MCS110+Carboplatin+Gemcitabine | MCS110 With C1D8 Dose + Carboplatin +Gemcitabine
Number analyzed (Participants) | 19 | 15
% change from baseline
  CD163: number analyzed (Participants) | 10 | 5
  CD163 | 42.1 (62.1) | 43.5 (239.5)
  CD8: number analyzed (Participants) | 9 | 5
  CD8 | 102 (747.3) | 99.0 (92.2)

13. Secondary Outcome: Circulating Monocytes Cells in Blood
Description: Cycle duration is 21 days results expressed in percentage of cells. Only 1 arm reported as results were available for 1 patient only.
Time Frame: day 15, 29, 43, 50
Population: safety set: only 1 patient with data collected
Measure: Number; unit: percentage
Arm/Group | MCS110+Carboplatin+Gemcitabine
Number analyzed (Participants) | 1
percentage
  day 15 CD14+CD16- | 43.5
  day 15 CD14+CD16+ | 54.8
  day 29 (cycle 2 day 8) CD14+CD16- | 86.6
  day 29 (cycle 2 day 8) CD14+CD16+ | 12.2
  day 43 (cycle 3 day 1) CD14+CD16- | 9.1
  day 43 (cycle 3 day 1) CD14+CD16+ | 89.7
  day 50 (cycle 3 day 8) CD14+CD16- | 86
  day 50 (cycle 3 day 8) CD14+CD16+ | 10

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study treatment until end of study treatment plus up to 150 days post treatment, up to maximum duration of 5 years
Groups:
- MCS110 + Carbo/Gem: MCS110 + Carbo/Gem
- MCS110 With C1D8@Dose + Carbo/Gem: MCS110 with C1D8@dose + Carbo/Gem
- All MCS110 + @Carbo/Gem Patients: All MCS110 + @Carbo/Gem Patients
- Carbo/Gem: Carbo/Gem
- All@Patients: All@Patients
Arm/Group | MCS110 + Carbo/Gem | MCS110 With C1D8@Dose + Carbo/Gem | All MCS110 + @Carbo/Gem Patients | Carbo/Gem | All@Patients
All-Cause Mortality (participants affected / at risk) | 1/19 | 1/15 | 2/34 | 1/15 | 3/49
Serious Adverse Events (participants affected / at risk) | 10/19 | 7/15 | 17/34 | 1/15 | 18/49
Other Adverse Events (participants affected / at risk) | 19/19 | 15/15 | 34/34 | 15/15 | 49/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MCS110 + Carbo/Gem (N=19) | MCS110 With C1D8@Dose + Carbo/Gem (N=15) | All MCS110 + @Carbo/Gem Patients (N=34) | Carbo/Gem (N=15) | All@Patients (N=49)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 1
Atypical haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 3 | 3 | 0 | 3
Myocardial ischaemia (Cardiac disorders) | 0 | 1 | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 1
Obstructive pancreatitis (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2 | 2 | 0 | 2
Fatigue (General disorders) | 0 | 1 | 1 | 0 | 1
Generalised oedema (General disorders) | 1 | 0 | 1 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 1 | 0 | 1
Device related infection (Infections and infestations) | 1 | 0 | 1 | 0 | 1
Erysipelas (Infections and infestations) | 1 | 0 | 1 | 0 | 1
Genital infection (Infections and infestations) | 1 | 0 | 1 | 0 | 1
Infection (Infections and infestations) | 0 | 1 | 1 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 1 | 0 | 1
Mastitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Sepsis (Infections and infestations) | 1 | 0 | 1 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 1 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 1 | 0 | 1
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1 | 1 | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 1 | 2 | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 3 | 0 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 1
Hypertension (Vascular disorders) | 1 | 0 | 1 | 0 | 1
Hypertensive crisis (Vascular disorders) | 0 | 1 | 1 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MCS110 + Carbo/Gem (N=19) | MCS110 With C1D8@Dose + Carbo/Gem (N=15) | All MCS110 + @Carbo/Gem Patients (N=34) | Carbo/Gem (N=15) | All@Patients (N=49)
Anaemia (Blood and lymphatic system disorders) | 13 | 10 | 23 | 10 | 33
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 5 | 6 | 3 | 9
Neutropenia (Blood and lymphatic system disorders) | 10 | 8 | 18 | 8 | 26
Thrombocytopenia (Blood and lymphatic system disorders) | 8 | 8 | 16 | 8 | 24
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 1 | 1 | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 0 | 1 | 0 | 1
Palpitations (Cardiac disorders) | 1 | 0 | 1 | 1 | 2
Tachycardia (Cardiac disorders) | 1 | 1 | 2 | 0 | 2
Vertigo (Ear and labyrinth disorders) | 1 | 1 | 2 | 0 | 2
Hypothyroidism (Endocrine disorders) | 2 | 0 | 2 | 0 | 2
Conjunctival haemorrhage (Eye disorders) | 0 | 1 | 1 | 0 | 1
Diplopia (Eye disorders) | 0 | 0 | 0 | 1 | 1
Dry eye (Eye disorders) | 1 | 0 | 1 | 0 | 1
Eye oedema (Eye disorders) | 0 | 1 | 1 | 0 | 1
Eye pain (Eye disorders) | 1 | 0 | 1 | 0 | 1
Eyelid oedema (Eye disorders) | 2 | 0 | 2 | 0 | 2
Foreign body sensation in eyes (Eye disorders) | 1 | 0 | 1 | 0 | 1
Lacrimation increased (Eye disorders) | 2 | 1 | 3 | 0 | 3
Orbital oedema (Eye disorders) | 0 | 1 | 1 | 0 | 1
Periorbital oedema (Eye disorders) | 8 | 6 | 14 | 0 | 14
Periorbital swelling (Eye disorders) | 1 | 0 | 1 | 0 | 1
Vision blurred (Eye disorders) | 1 | 1 | 2 | 0 | 2
Xerophthalmia (Eye disorders) | 0 | 0 | 0 | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 4 | 3 | 7 | 1 | 8
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1 | 3 | 0 | 3
Chapped lips (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 5 | 3 | 8 | 2 | 10
Diarrhoea (Gastrointestinal disorders) | 5 | 2 | 7 | 3 | 10
Dry mouth (Gastrointestinal disorders) | 2 | 0 | 2 | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 2 | 1 | 3 | 3 | 6
Flatulence (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 1
Gingival bleeding (Gastrointestinal disorders) | 1 | 1 | 2 | 0 | 2
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Gingival recession (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1
Lip oedema (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 10 | 12 | 22 | 8 | 30
Odynophagia (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 1
Periodontal disease (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 2
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1
Salivary hypersecretion (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 2 | 5 | 7 | 1 | 8
Vomiting (Gastrointestinal disorders) | 5 | 3 | 8 | 2 | 10
Asthenia (General disorders) | 5 | 3 | 8 | 4 | 12
Chest discomfort (General disorders) | 0 | 1 | 1 | 0 | 1
Chills (General disorders) | 2 | 2 | 4 | 0 | 4
Device related thrombosis (General disorders) | 0 | 0 | 0 | 1 | 1
Face oedema (General disorders) | 4 | 3 | 7 | 0 | 7
Facial pain (General disorders) | 1 | 0 | 1 | 0 | 1
Fatigue (General disorders) | 6 | 9 | 15 | 4 | 19
Gait disturbance (General disorders) | 0 | 1 | 1 | 0 | 1
General physical health deterioration (General disorders) | 1 | 0 | 1 | 0 | 1
Influenza like illness (General disorders) | 0 | 1 | 1 | 1 | 2
Infusion site extravasation (General disorders) | 0 | 0 | 0 | 1 | 1
Infusion site pain (General disorders) | 0 | 1 | 1 | 0 | 1
Injection site reaction (General disorders) | 0 | 1 | 1 | 0 | 1
Injection site swelling (General disorders) | 0 | 1 | 1 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1 | 1
Oedema peripheral (General disorders) | 3 | 4 | 7 | 1 | 8
Peripheral swelling (General disorders) | 1 | 1 | 2 | 0 | 2
Pyrexia (General disorders) | 4 | 3 | 7 | 2 | 9
Swelling (General disorders) | 1 | 0 | 1 | 0 | 1
Swelling face (General disorders) | 2 | 0 | 2 | 0 | 2
Xerosis (General disorders) | 0 | 0 | 0 | 1 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 1 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1 | 1 | 2 | 3
Bronchitis viral (Infections and infestations) | 1 | 0 | 1 | 0 | 1
Candida infection (Infections and infestations) | 1 | 0 | 1 | 0 | 1
Catheter site infection (Infections and infestations) | 1 | 0 | 1 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Cystitis (Infections and infestations) | 1 | 0 | 1 | 0 | 1
Ear infection (Infections and infestations) | 1 | 0 | 1 | 0 | 1
Folliculitis (Infections and infestations) | 1 | 0 | 1 | 0 | 1
Fungal oesophagitis (Infections and infestations) | 1 | 0 | 1 | 0 | 1
Gingivitis (Infections and infestations) | 1 | 0 | 1 | 0 | 1
Influenza (Infections and infestations) | 1 | 0 | 1 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 0 | 1
Lymphangitis (Infections and infestations) | 1 | 0 | 1 | 0 | 1
Mastitis (Infections and infestations) | 1 | 0 | 1 | 0 | 1
Nail infection (Infections and infestations) | 1 | 0 | 1 | 0 | 1
Oral candidiasis (Infections and infestations) | 1 | 0 | 1 | 1 | 2
Oral herpes (Infections and infestations) | 1 | 1 | 2 | 2 | 4
Oral infection (Infections and infestations) | 1 | 0 | 1 | 0 | 1
Oropharyngeal candidiasis (Infections and infestations) | 1 | 0 | 1 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 2 | 2 | 0 | 2
Sinusitis (Infections and infestations) | 0 | 1 | 1 | 1 | 2
Spinal cord infection (Infections and infestations) | 1 | 0 | 1 | 0 | 1
Tinea pedis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Tonsillitis (Infections and infestations) | 0 | 1 | 1 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 2 | 3 | 2 | 5
Urinary tract infection (Infections and infestations) | 1 | 2 | 3 | 0 | 3
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 1
Chemical cystitis (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 2 | 1 | 3 | 1 | 4
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Oral contusion (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 1
Seroma (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 1
Alanine aminotransferase increased (Investigations) | 12 | 12 | 24 | 2 | 26
Amylase increased (Investigations) | 1 | 1 | 2 | 0 | 2
Aspartate aminotransferase increased (Investigations) | 16 | 12 | 28 | 4 | 32
Blood alkaline phosphatase increased (Investigations) | 4 | 1 | 5 | 0 | 5
Blood creatine phosphokinase MB increased (Investigations) | 1 | 0 | 1 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 9 | 7 | 16 | 0 | 16
Blood creatinine increased (Investigations) | 1 | 2 | 3 | 0 | 3
Blood iron decreased (Investigations) | 0 | 0 | 0 | 1 | 1
Blood lactate dehydrogenase increased (Investigations) | 2 | 1 | 3 | 0 | 3
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 1 | 1
Gamma-glutamyltransferase increased (Investigations) | 5 | 1 | 6 | 0 | 6
Haemoglobin decreased (Investigations) | 1 | 1 | 2 | 0 | 2
Hepatic enzyme increased (Investigations) | 1 | 0 | 1 | 0 | 1
Lipase (Investigations) | 1 | 0 | 1 | 0 | 1
Lipase increased (Investigations) | 0 | 1 | 1 | 0 | 1
Lymphocyte count decreased (Investigations) | 2 | 1 | 3 | 0 | 3
Neutrophil count decreased (Investigations) | 6 | 5 | 11 | 5 | 16
Platelet count decreased (Investigations) | 3 | 3 | 6 | 6 | 12
Weight decreased (Investigations) | 1 | 1 | 2 | 0 | 2
Weight increased (Investigations) | 0 | 2 | 2 | 0 | 2
White blood cell count decreased (Investigations) | 3 | 4 | 7 | 1 | 8
Decreased appetite (Metabolism and nutrition disorders) | 3 | 4 | 7 | 2 | 9
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 1
Fluid retention (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 0 | 2 | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 1 | 2 | 0 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 0 | 2 | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1 | 3 | 0 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 1 | 3 | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2 | 1 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 2 | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 1
Fracture pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 1 | 4 | 1 | 5
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1 | 3 | 0 | 3
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 1
Ageusia (Nervous system disorders) | 1 | 0 | 1 | 0 | 1
Balance disorder (Nervous system disorders) | 1 | 0 | 1 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 2 | 2 | 0 | 2
Dysaesthesia (Nervous system disorders) | 0 | 1 | 1 | 0 | 1
Dysgeusia (Nervous system disorders) | 1 | 1 | 2 | 0 | 2
Headache (Nervous system disorders) | 4 | 3 | 7 | 4 | 11
Myelopathy (Nervous system disorders) | 0 | 1 | 1 | 0 | 1
Neuralgia (Nervous system disorders) | 2 | 0 | 2 | 0 | 2
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 1 | 1 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 3 | 3 | 1 | 4
Vocal cord paralysis (Nervous system disorders) | 1 | 0 | 1 | 0 | 1
Device dislocation (Product Issues) | 0 | 1 | 1 | 0 | 1
Anxiety (Psychiatric disorders) | 2 | 2 | 4 | 1 | 5
Depressed mood (Psychiatric disorders) | 1 | 1 | 2 | 0 | 2
Depression (Psychiatric disorders) | 1 | 0 | 1 | 2 | 3
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1
Insomnia (Psychiatric disorders) | 1 | 0 | 1 | 1 | 2
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1
Nocturia (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 1
Breast oedema (Reproductive system and breast disorders) | 0 | 1 | 1 | 0 | 1
Breast pain (Reproductive system and breast disorders) | 1 | 2 | 3 | 0 | 3
Menorrhagia (Reproductive system and breast disorders) | 1 | 0 | 1 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 1 | 0 | 1 | 0 | 1
Aphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 1
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 7 | 0 | 7
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 3 | 0 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 5 | 11 | 2 | 13
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 4 | 0 | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 1
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2 | 0 | 2
Snoring (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 1
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 2 | 3 | 3 | 6
Blood blister (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 3 | 3 | 0 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 2 | 4 | 0 | 4
Erythema (Skin and subcutaneous tissue disorders) | 0 | 3 | 3 | 0 | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 3 | 5 | 0 | 5
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 5 | 5 | 10 | 4 | 14
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 0 | 2
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 1
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 1
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 1
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 1
Flushing (Vascular disorders) | 1 | 0 | 1 | 1 | 2
Haematoma (Vascular disorders) | 1 | 0 | 1 | 0 | 1
Hot flush (Vascular disorders) | 0 | 0 | 0 | 1 | 1
Hypertension (Vascular disorders) | 3 | 1 | 4 | 0 | 4
Hypotension (Vascular disorders) | 1 | 0 | 1 | 0 | 1
Jugular vein thrombosis (Vascular disorders) | 1 | 0 | 1 | 0 | 1
Peripheral venous disease (Vascular disorders) | 0 | 0 | 0 | 1 | 1
Phlebitis (Vascular disorders) | 0 | 1 | 1 | 0 | 1
Poor venous access (Vascular disorders) | 0 | 0 | 0 | 1 | 1
Thrombophlebitis (Vascular disorders) | 0 | 0 | 0 | 2 | 2
Thrombosis (Vascular disorders) | 1 | 0 | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-10-11): https://cdn.clinicaltrials.gov/large-docs/80/NCT02435680/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-29): https://cdn.clinicaltrials.gov/large-docs/80/NCT02435680/SAP_001.pdf